CLINICAL TRIAL: NCT01651949
Title: A Phase III Clinical Trial to Study the Tolerability and Immunogenicity of 9vHPV (V503), a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine, in 16- to 26-Year-Old Men and 16- to 26-Year-Old Women
Brief Title: Multivalent HPV (Human Papillomavirus) Vaccine Study in 16- to 26-Year Old Men and Women (V503-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-003; 2012-002758-22 (EudraCT Number)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Genital Warts; Anal Cancer; Anal Intraepithelial Neoplasia
MeSH Terms: conditions — Condylomata Acuminata; Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Females (Active Comparator): Healthy females 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: 9vHPV Vaccine
- Heterosexual Males (Experimental): Healthy heterosexual males 16 to 26 years of age received 9vHPV 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: 9vHPV Vaccine
- Men who have Sex with Men (Experimental): Healthy MSM 16 to 26 years of age received 9vHPV 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: 9vHPV Vaccine

INTERVENTIONS:
Biological: 9vHPV Vaccine — 9vHPV, V503 (9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine), 0.5 mL injection in 3-dose regimen

SUMMARY:
This study is designed to evaluate the immunogenicity and tolerability of 9vHPV (9-valent HPV vaccine, V503) in 16- to 26-year old men and women. The overall goal is to bridge 9vHPV efficacy findings in young women to young men based on the demonstration of similar immunogenicity and safety profiles. The primary hypothesis is that 9vHPV induces antibody responses at 4 weeks postdose 3 in heterosexual males that are non-inferior to antibody responses in young women.

DETAILED DESCRIPTION:
Study participants will be administered a 3-dose regimen of 9vHPV. They will be assessed for immunogenicity 1 month following completion of vaccination. All participants will be followed for safety for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Good physical health
* Has never had Papanicolaou testing (Pap, cervical or anal) or has only had normal Pap test results
* Other inclusion criteria will be discussed with the investigator

Exclusion Criteria:

* History of severe allergic reaction that required medical intervention
* Currently enrolled in a clinical trial
* If participant is female, pregnant
* Currently immunocompromised or having received immunosuppressive therapy in the last year
* Positive test for HPV
* History of HPV-related external genital lesions or HPV-related anal lesions or anal cancer
* If participant is female, history of abnormal cervical biopsy results
* Other exclusion criteria will be discussed with the investigator

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2520 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2014-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Castellsague X, Giuliano AR, Goldstone S, Guevara A, Mogensen O, Palefsky JM, Group T, Shields C, Liu K, Maansson R, Luxembourg A, Kaplan SS. Immunogenicity and safety of the 9-valent HPV vaccine in men. Vaccine. 2015 Nov 27;33(48):6892-901. doi: 10.1016/j.vaccine.2015.06.088. Epub 2015 Jul 2. PMID 26144901
- [Derived] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-003&kw=V503-003&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Heterosexual Males: Healthy heterosexual males 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
- Females: Healthy females 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
- Men Who Have Sex With Men (MSM): Healthy MSM 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
Period: Overall Study
Arm/Group | Heterosexual Males | Females | Men Who Have Sex With Men (MSM)
Started | 1106 | 1101 | 313
Vaccination 1 | 1103 | 1099 | 313
Vaccination 2 | 1089 | 1069 | 298
Vaccination 3 | 1067 | 1037 | 291
Completed | 1053 | 1015 | 282
Not Completed | 53 | 86 | 31
Not completed — Unknown status | 4 | 4 | 0
Not completed — Lost to Follow-up | 30 | 56 | 20
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Screen failure | 2 | 2 | 0
Not completed — Withdrawal by Subject | 17 | 18 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heterosexual Males | Females | Men Who Have Sex With Men (MSM) | Total
Number analyzed (Participants) | 1106 | 1101 | 313 | 2520
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (3.0) | 21.3 (2.9) | 22.2 (2.4) | 21.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1101 | 0 | 1101
  Male | 1106 | 0 | 313 | 1419

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) to the HPV Types Contained in the 9vHPV Vaccine
Description: Serum antibodies to HPV types 6/11/16/18/31/33/45/52/58 were measured with a Competitive Luminex Immunoassay. Titers are reported in milli Merck Units/mL
Time Frame: Four weeks post vaccination 3 (Month 7)
Population: The analysis set includes heterosexual male and female participants who received the 3 vaccinations, were seronegative to the appropriate HPV type at baseline, and had Month 7 immunogenicity results for the appropriate HPV type. Per-protocol non-inferiority analysis compared heterosexual males and females only.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Groups:
- Men Who Have Sex With Men: Healthy MSM 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
Arm/Group | Heterosexual Males | Females | Men Who Have Sex With Men
Number analyzed (Participants) | 914 | 884 | 239
milli Merck Units/mL
  Anti-HPV Type 6 (n=847, 708, 164) | 782.0 [738.0 to 828.7] | 703.9 [660.6 to 749.9] | 568.9 [498.7 to 649.0]
  Anti-HPV Type 11 (n=851, 712, 165) | 616.7 [582.4 to 653.0] | 564.9 [530.6 to 601.3] | 437.7 [384.4 to 498.5]
  Anti-HPV Type 16 (n=899, 781, 212) | 3346.0 [3158.9 to 3544.1] | 2788.3 [2621.4 to 2965.8] | 2294.0 [2037.8 to 2582.5]
  Anti-HPV Type 18 (n=906, 831, 220) | 808.2 [754.9 to 865.4] | 679.8 [633.1 to 730.1] | 608.1 [529.4 to 698.5]
  Anti-HPV Type 31 (n=908, 826, 227) | 708.5 [662.7 to 757.6] | 570.1 [531.5 to 611.5] | 420.7 [368.0 to 480.9]
  Anti-HPV Type 33 (n=901, 853, 230) | 384.8 [362.5 to 408.4] | 322.0 [302.9 to 342.3] | 252.3 [224.2 to 283.8]
  Anti-HPV Type 45 (n=909, 871, 232) | 235.6 [219.0 to 253.6] | 185.7 [172.3 to 200.2] | 157.5 [136.2 to 182.2]
  Anti-HPV Type 52 (n=907, 849, 232) | 386.8 [363.4 to 411.6] | 335.2 [314.3 to 357.6] | 233.1 [206.0 to 263.7]
  Anti-HPV Type 58 (n=897, 839, 223) | 509.8 [479.9 to 541.6] | 409.3 [384.5 to 435.7] | 319.8 [283.2 to 361.0]
Statistical Analysis 1: Comparison: Heterosexual Males vs Females; Anti-HPV Type 6; Test type: Non-Inferiority or Equivalence — Criterion for non-inferiority with respect to GMT ratio (heterosexual males / females) required that the lower bound of the 95% confidence interval was >0.67, to exclude a decrease of 1.5-fold or more; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.11, 95% CI 2-sided [1.02 to 1.21]
Statistical Analysis 2: Comparison: Heterosexual Males vs Females; Anti-HPV Type 11; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.09, 95% CI 2-sided [1.00 to 1.19]
Statistical Analysis 3: Comparison: Heterosexual Males vs Females; Anti-HPV Type 16; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.20, 95% CI 2-sided [1.10 to 1.30]
Statistical Analysis 4: Comparison: Heterosexual Males vs Females; Anti-HPV Type 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.19, 95% CI 2-sided [1.08 to 1.31]
Statistical Analysis 5: Comparison: Heterosexual Males vs Females; Anti-HPV Type 31; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.24, 95% CI 2-sided [1.13 to 1.37]
Statistical Analysis 6: Comparison: Heterosexual Males vs Females; Anti-HPV Type 33; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.19, 95% CI 2-sided [1.10 to 1.30]
Statistical Analysis 7: Comparison: Heterosexual Males vs Females; Anti-HPV Type 45; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.27, 95% CI 2-sided [1.14 to 1.41]
Statistical Analysis 8: Comparison: Heterosexual Males vs Females; Anti-HPV Type 52; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.15, 95% CI 2-sided [1.05 to 1.26]
Statistical Analysis 9: Comparison: Heterosexual Males vs Females; Anti-HPV Type 58; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; An analysis of variance model with a response of log individual titers and fixed effect for group was used; GMT Ratio = 1.25, 95% CI 2-sided [1.14 to 1.36]

2. Primary Outcome: Percentage of Participants With One or More Injection-site Adverse Experiences Prompted on the Vaccination Report Card
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Injection-site AEs prompted on the Vaccination Report Card (VRC) were erythema, pain, and swelling. Participants were instructed to use the Vaccination Report Card to record AEs daily after each study vaccination.
Time Frame: Up to 5 days after any vaccination
Population: The analysis set includes all participants who received >=1 vaccination and had safety follow-up. Heterosexual and MSM males were combined for safety outcomes.
Measure: Number; unit: Percentage of Participants
Groups:
- Heterosexual and MSM Males: Healthy heterosexual and MSM males 16 to 26 years of age received 9vHPV vaccine 0.5 mL intramuscular injection on Day 1, Month 1, and Month 6
Arm/Group | Heterosexual and MSM Males | Females
Number analyzed (Participants) | 1394 | 1075
Percentage of Participants
  Overall injection-site AEs | 66.7 | 84.0
  Injection-site Erythema | 20.7 | 32.2
  Injection-site Pain | 63.4 | 82.5
  Injection-site Swelling | 20.2 | 37.5
Statistical Analysis 1: Comparison: Heterosexual and MSM Males vs Females; Injection-site Erythema; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = -11.5, 95% CI 2-sided [-15.0 to -8.0] — The incidence of AEs of injection-site erythema reported on the Vaccination Report Card was compared between heterosexual / MSM male participants and female participants
Statistical Analysis 2: Comparison: Heterosexual and MSM Males vs Females; Injection-site Pain; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = -19.1, 95% CI 2-sided [-22.5 to -15.7] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Heterosexual and MSM Males vs Females; Injection-site Swelling; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = -17.3, 95% CI 2-sided [-20.8 to -13.7] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Percentage of Participants With Elevated Oral Body Temperature (>=37.8° C, >=100° F)
Description: Participants were instructed by the investigator to use the Vaccination Report Card to document evening oral temperature daily after each study vaccination
Time Frame: Up to 5 days after any vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Heterosexual and MSM Males | Females
Number analyzed (Participants) | 1386 | 1066
Percentage of Participants | 4.4 | 5.9
Statistical Analysis 1: Comparison: Heterosexual and MSM Males vs Females; Elevated Body Temperature; Test type: Superiority or Other; p = 0.091, Miettinen & Nurminen; Risk Difference (RD) = -1.5, 95% CI 2-sided [-3.4 to 0.2] — The incidence of maximum body temperature >=37.8° C reported on the Vaccination Report Card was compared between heterosexual / MSM male participants and female participants

4. Secondary Outcome: Percentage of Participants With Seroconversion to the HPV Types Contained in the 9vHPV Vaccine
Description: Serum antibodies to HPV types were measured with a Competitive Luminex Immunoassay. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30; HPV Type 11: ≥16; HPV Type 16: ≥20; HPV Type 18: ≥24; HPV Type 31: ≥10; HPV Types 33, 45, 52, and 58: ≥8.
Time Frame: Four weeks post vaccination 3 (Month 7)
Population: The analysis set includes participants who received the 3 vaccinations, were seronegative to the appropriate HPV type at baseline, and had Month 7 immunogenicity results for the appropriate HPV type. Per-protocol non-inferiority analysis compared heterosexual males and females only.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Heterosexual Males | Females | Men Who Have Sex With Men
Number analyzed (Participants) | 914 | 884 | 239
Percentage of Participants
  Anti-HPV Type 6 (n=847, 708, 164) | 99.6 [99.0 to 99.9] | 99.6 [98.8 to 99.9] | 99.4 [96.6 to 100]
  Anti-HPV Type 11 (n=851, 712, 165) | 100 [99.6 to 100] | 99.9 [99.2 to 100] | 100 [97.8 to 100]
  Anti-HPV Type 16 (n=899, 781, 212) | 100 [99.6 to 100] | 99.9 [99.3 to 100] | 100 [98.3 to 100]
  Anti-HPV Type 18 (n=906, 831, 220) | 99.9 [99.4 to 100] | 99.8 [99.1 to 100] | 99.5 [97.5 to 100]
  Anti-HPV Type 31 (n=908, 826, 227) | 100 [99.6 to 100] | 100 [99.6 to 100] | 100 [98.4 to 100]
  Anti-HPV Type 33 (n=901, 853, 230) | 100 [99.6 to 100] | 99.9 [99.3 to 100] | 100 [98.4 to 100]
  Anti-HPV Type 45 (n=909, 871, 232) | 99.8 [99.2 to 100] | 99.5 [98.8 to 99.9] | 100 [98.4 to 100]
  Anti-HPV Type 52 (n=907, 849, 232) | 100 [99.6 to 100] | 99.8 [99.2 to 100] | 100 [98.4 to 100]
  Anti-HPV Type 58 (n=897, 839, 223) | 100 [99.6 to 100] | 99.8 [99.1 to 100] | 100 [98.4 to 100]
Statistical Analysis 1: Comparison: Heterosexual Males vs Females; Anti-HPV Type 6; Test type: Non-Inferiority or Equivalence — Criterion for non-inferiority with respect to seroconversion percentage (heterosexual males minus females) required that the lower bound of the 95% confidence interval was greater than -5; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.7 to 0.9]
Statistical Analysis 2: Comparison: Heterosexual Males vs Females; Anti-HPV Type 11; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.3 to 0.8]
Statistical Analysis 3: Comparison: Heterosexual Males vs Females; Anti-HPV Type 16; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 4: Comparison: Heterosexual Males vs Females; Anti-HPV Type 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.4 to 0.8]
Statistical Analysis 5: Comparison: Heterosexual Males vs Females; Anti-HPV Type 31; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.0, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 6: Comparison: Heterosexual Males vs Females; Anti-HPV Type 33; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 7: Comparison: Heterosexual Males vs Females; Anti-HPV Type 45; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.2, 95% CI 2-sided [-0.4 to 1.0]
Statistical Analysis 8: Comparison: Heterosexual Males vs Females; Anti-HPV Type 52; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.2, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 9: Comparison: Heterosexual Males vs Females; Anti-HPV Type 58; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 0.2, 95% CI 2-sided [-0.2 to 0.9]

5. Primary Outcome: Percentage of Participants With an Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE.
Time Frame: Up to Month 12
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Heterosexual and MSM Males | Females
Number analyzed (Participants) | 1394 | 1075
Percentage of Participants | 76.2 | 89.4

6. Primary Outcome: Percentage of Participants Who Had Study Vaccine Discontinued Due to an Adverse Event
Description: as for outcome 5
Time Frame: Up to Month 12
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Heterosexual and MSM Males | Females
Number analyzed (Participants) | 1394 | 1075
Percentage of Participants | 0.1 | 0.3

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: The analysis set includes all participants who received >=1 vaccination and had safety follow-up. Heterosexual and MSM males were combined for safety outcomes.
Arm/Group | Heterosexual and MSM Males | Females
Serious Adverse Events (participants affected / at risk) | 23/1394 | 26/1075
Other Adverse Events (participants affected / at risk) | 976/1394 | 924/1075
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heterosexual and MSM Males (N=1394) | Females (N=1075)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Familial periodic paralysis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cyst rupture (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
External ear cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophreniform disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 4 (4)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heterosexual and MSM Males (N=1394) | Females (N=1075)
Injection site erythema (General disorders) | 291 (422) | 348 (539)
Injection site pain (General disorders) | 886 (1877) | 893 (2101)
Injection site swelling (General disorders) | 285 (431) | 408 (661)
Headache (Nervous system disorders) | 200 (271) | 246 (378)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.